CLINICAL TRIAL: NCT06939257
Title: The Impact of Gender Affirming Hormone Therapy on Pain In Gender Minority Adults
Acronym: TRANSPIRE
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00160765; 1R01NS135833-01A1 (NIH)
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pain; Gender Minority Individuals
Keywords: GHT; Gender Minority; HRT; Gender Affirming Hormone Therapy; GM
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples may be retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons Initiating GHT
- Gender Minority Persons Not Taking GHT

SUMMARY:
TRANSPIRE is an observational study of ~200 individuals who (1) will be initiating gender-affirming hormone therapy (GHT) or (2) are gender minority individuals who do not use GHT. The primary outcome will be to identify how the presence of chronic pain changes overtime with GHT through the use of surveys, quantitative sensory testing (QST), brain MRIs, and qualitative interviews.

Following recruitment and consent, participants will complete baseline survey measures and will repeat those measures at 1 months, 3 month, 6 months, and 12 months. QST measures, brain MRIs, and Qualitative Interviews will be offered to participants in cohort (1) and will be completed at baseline and 12 months.

DETAILED DESCRIPTION:
In most chronic pain syndromes there is a 1.5-2 times higher incidence in females compared to males after puberty, which may in part be due to differences in sex hormone levels and receptors and/or other unknown mechanisms related to sex and/or gender. Gender-affirming hormone therapy (GHT) is routinely used in gender minority (GM) persons' gender-affirming medical care. Masculinizing GHT includes the use of testosterone, whereas feminizing GHT includes estrogen and progesterone, often in conjunction with an anti- androgen. In 2011, The Institute of Medicine identified GM adults as an understudied population in critical need of more health-related research. The GM community includes those who identify as transgender men (TGM), transgender women (TGW), and as non-binary (persons whose gender is not binary). There are only a few studies on how GHT is related to the presence and severity of pain in GM persons. Previous research has shown that GM persons have been reported to have an overall greater prevalence of multiple chronic pain syndromes compared to cisgender persons (persons whose gender corresponds to their sex assigned at birth). Retrospective and cross-sectional studies have identified that GHT may affect the presence and severity of chronic pain in the GM population, with masculinizing GHT being potentially associated with improvements in chronic pain and feminizing GHT with estrogen/progesterone and anti-androgens potentially worsening chronic pain. Investigators hypothesize that the presence of androgenic hormonal influences is protective against the development of a specific chronic pain mechanism, nociplastic pain - pain that appears to be driven by the central nervous system (CNS). The mechanisms that underlie nociplastic pain are not entirely understood, but it is thought that amplified and/or dysregulated pain and sensory signaling within the CNS plays a substantial role. Numerous chronic pain syndromes have been identified as primarily nociplastic and include fibromyalgia, tension headache, and chronic low back pain. These and other pain syndromes often co-occur and are recognized by the NIH as Chronic Overlapping Pain Conditions (COPCs). A large knowledge gap exists and thus presents a unique opportunity to study how GHT may influence the presence and severity of pain in GM persons using a rigorous longitudinal design.

Aim 1: To characterize the trajectory of pain and pain-related symptoms in GM adults taking GHT.

Aim 2: To perform quantitative sensory testing (QST) and functional brain neuroimaging of GM adults undergoing GHT to examine the mechanism(s) that underlie changes in pain and sensory sensitivity associated with GHT.

Aim 3: To perform qualitative studies of how GHT affects gender affirmation, psychological wellbeing, and the experience of pain. Investigators will perform and communicate results of these studies using a community-engaged approach.

Data from our work will better enable clinicians to inform GM patients about potential pain-related changes that may occur with GHT and support future studies on mechanisms-based interventions to treat and mitigate chronic pain during gender-affirming care.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the participant
* Ages 18-50 years
* English speaking
* GM persons who have been deemed to be an appropriate medical candidate to take gender-affirming hormone therapy for gender incongruence -OR- GM persons who are not taking gender-affirming hormone therapy

Aim 2 (QST and MRI) Additional Inclusion Criteria:

* GM persons who have been deemed to be an appropriate medical candidate to take gender- affirming hormone therapy for gender incongruence
* Stable doses of analgesic medications for at least 30 days prior to screening
* Right handed
* Normal visual acuity or correctable to at least 20/40 for reading instructions in the MRI
* Willingness to refrain from pain medications such as NSAIDs, acetaminophen, and opioid medications for 12 hours prior to neuroimaging and QST
* Willingness to refrain from alcohol and nicotine on day of QST and neuroimaging
* Willingness to refrain from physical activity or exercise that would cause muscle and/or joint soreness for 48 hours prior to testing (routine exercise or activity that does not lead to soreness is acceptable)
* Investigators will attempt to recruit individuals with no chronic daily use of adjunctive pain medications, including tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors, and gabapentinoids as these drugs can influence neuroimaging and QST findings, or have individuals be weaned off of these meds at least two weeks prior to being studied. In previous smaller imaging studies investigators could accomplish this, but this may not be possible in this large of a study. If the study team does need to allow individuals into these cohorts while on such medications because of pragmatic issues, this information will be recorded and patients will be asked to remain on a stable dose for at least two weeks prior to MRI and QST assessments.
* Able to lie still on their back for 1.5 hours for MRI scans

Exclusion Criteria:

* Inability to provide informed consent
* Age less than 18 years or greater than 50 years
* Severe physical impairment (e.g., blindness, deafness, paraplegia)
* Co-morbid medical conditions that may significantly impair physical functional status (e.g., history of non-skin malignancy, or autoimmune disorder)
* Pregnant or nursing
* Liver failure
* Self-reported liver cirrhosis
* Self-reported hepatitis
* Severe Cardiovascular disease (examples: history of myocardial infarction, unstable angina, severe coronary artery disease, congestive heart failure, or severe valvular abnormalities) that are self-reported by patient or by medical record
* Prisoner
* Current litigation for chronic pain
* Current disability proceedings
* Active psychotic or suicidal symptoms
* Current drug or alcohol use disorder
* History of gonadectomy surgery

Aim 2 (QST and MRI) Additional Inclusion Criteria:

* Contraindications to MRI (e.g., metal implants, pacemaker, etc.)
* Severe claustrophobia precluding MRI and evoked pain testing during scanning
* BMI > 40 or unable to lie comfortably in MRI
* Current, recent (within the last 6 months), or habitual use of artificial nails or nail enhancements. (Artificial nails can influence pressure pain sensitivity at the thumbnail)
* Peripheral neuropathy
* Diagnosed epilepsy or seizure history

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All gender minority persons
Study Population: Gender minority individuals from within the greater Kansas City area
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2029-09-16 (Estimated); Study Completion 2029-09-16 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Chronic Pain in Gender Minority Adults Initiating GHT | Baseline and 1, 3, 6, and 12-months.
  The primary outcome is to measure the presence of chronic pain before and after the initiation of GHT. Participants will be asked if they have had pain on more than half the days of the last 3 months.
fMRI Changes in Functional Connectivity | Baseline (pre-GHT) and 12-months (post-GHT)
  For Aim 2 (QST and MRI), the primary outcome is to identify changes in resting state functional connectivity (e.g., ACC - PAG) over time with GHT in GM persons on masculinizing GHT and GM persons on feminizing GHT.
Qualitative Interview Outcome Measure | Baseline (pre-GHT) and 12-month (post-GHT)
  1) To better understand the relationship between stress, loneliness, medical mistrust, affirmation treatment, chronic pain, and psychological functioning in GM persons. 2) To better understand the lived experiences of GM persons with and without chronic pain. 3) To better understand the lived experiences of GM persons and how gender-affirming care has impacted their overall physical and mental wellbeing.

SECONDARY OUTCOMES:
Severity of Chronic Pain | Baseline and 1, 3, 6, and 12-months
  For those GM participants with the presence of chronic pain, investigators will assess how pain severity NRS ratings change over time with GHT. This will be assessed using the Brief Pain Inventory (BPI) which assesses pain on a scale of 0-10 at its worst in the past 7 days, on average in the past 7 days, at its least in the past 7 days, and at the current time.
Magnitude of Nociplastic Pain | Baseline and 1, 3, 6, and 12-months.
  Investigators will use the 2016 Fibromyalgia Survey to assess the magnitude of pain. The 2016 FM survey consists of a body map score and Symptom Severity Index score that are added together to indicate the severity of Fibromyalgia. The higher the score, the higher the severity.
Quantitative Sensory Testing within the fMRI | Baseline (pre-GHT) and 12-months (post-GHT)
  For Aim 2, the secondary outcomes will be to identify changes in QST parameters before and after GHT-initiation. Two QST measures will be completed during each fMRI scan and values will be compared. Brain activation during the painful QST sensations will be measured and compared between the two time points.
Gray Matter Volume after initiating GHT | Baseline (pre-GHT) and 12-months (post-GHT)
  For Aim 2, gray matter may impact nerves and pain reception. The volume will be measured within the fMRI before and after initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Chadwick, MD, MSc, FASA, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartley EJ, King CD, Sibille KT, Cruz-Almeida Y, Riley JL 3rd, Glover TL, Goodin BR, Sotolongo AS, Herbert MS, Bulls HW, Staud R, Fessler BJ, Redden DT, Bradley LA, Fillingim RB. Enhanced Pain Sensitivity Among Individuals With Symptomatic Knee Osteoarthritis: Potential Sex Differences in Central Sensitization. Arthritis Care Res (Hoboken). 2016 Apr;68(4):472-80. doi: 10.1002/acr.22712. PMID 26434740
- [Background] Robinson ME, Wise EA, Gagnon C, Fillingim RB, Price DD. Influences of gender role and anxiety on sex differences in temporal summation of pain. J Pain. 2004 Mar;5(2):77-82. doi: 10.1016/j.jpain.2003.11.004. PMID 15042515
- [Background] Sarlani E, Grace EG, Reynolds MA, Greenspan JD. Sex differences in temporal summation of pain and aftersensations following repetitive noxious mechanical stimulation. Pain. 2004 May;109(1-2):115-23. doi: 10.1016/j.pain.2004.01.019. PMID 15082133
- [Background] Popescu A, LeResche L, Truelove EL, Drangsholt MT. Gender differences in pain modulation by diffuse noxious inhibitory controls: a systematic review. Pain. 2010 Aug;150(2):309-318. doi: 10.1016/j.pain.2010.05.013. Epub 2010 Jun 16. PMID 20557999
- [Background] Bulls HW, Freeman EL, Anderson AJ, Robbins MT, Ness TJ, Goodin BR. Sex differences in experimental measures of pain sensitivity and endogenous pain inhibition. J Pain Res. 2015 Jun 29;8:311-20. doi: 10.2147/JPR.S84607. eCollection 2015. PMID 26170713
- [Background] Mills SEE, Nicolson KP, Smith BH. Chronic pain: a review of its epidemiology and associated factors in population-based studies. Br J Anaesth. 2019 Aug;123(2):e273-e283. doi: 10.1016/j.bja.2019.03.023. Epub 2019 May 10. PMID 31079836
- [Background] Foxen-Craft E, Bourchtein E, Kaplan C, Clauw DJ, Scott E. Pain Widespreadedness, and Not Primary Pain Location, is Associated With Comorbid Symptoms in Children With Chronic Pain. Clin J Pain. 2023 Jan 1;39(1):1-7. doi: 10.1097/AJP.0000000000001083. PMID 36524767
- [Background] Abou L, Whibley D, Clauw DJ, Kratz AL. Widespread Pain With Nociplastic Features is an Independent Predictor of Low Physical Activity in People with Multiple Sclerosis. J Pain. 2024 Feb;25(2):418-427. doi: 10.1016/j.jpain.2023.09.005. Epub 2023 Sep 21. PMID 37741524
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Nijs J, Malfliet A, Nishigami T. Nociplastic pain and central sensitization in patients with chronic pain conditions: a terminology update for clinicians. Braz J Phys Ther. 2023 May-Jun;27(3):100518. doi: 10.1016/j.bjpt.2023.100518. Epub 2023 Jun 14. No abstract available. PMID 37348359
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Maixner W, Fillingim RB, Williams DA, Smith SB, Slade GD. Overlapping Chronic Pain Conditions: Implications for Diagnosis and Classification. J Pain. 2016 Sep;17(9 Suppl):T93-T107. doi: 10.1016/j.jpain.2016.06.002. PMID 27586833
- [Background] Kosek E, Clauw D, Nijs J, Baron R, Gilron I, Harris RE, Mico JA, Rice ASC, Sterling M. Chronic nociplastic pain affecting the musculoskeletal system: clinical criteria and grading system. Pain. 2021 Nov 1;162(11):2629-2634. doi: 10.1097/j.pain.0000000000002324. No abstract available. PMID 33974577
- [Background] Bazzichi L, Giacomelli C, Consensi A, Giorgi V, Batticciotto A, Di Franco M, Sarzi-Puttini P. One year in review 2020: fibromyalgia. Clin Exp Rheumatol. 2020 Jan-Feb;38 Suppl 123(1):3-8. Epub 2020 Feb 21. PMID 32116216
- [Background] Fitzcharles MA, Cohen SP, Clauw DJ, Littlejohn G, Usui C, Hauser W. Nociplastic pain: towards an understanding of prevalent pain conditions. Lancet. 2021 May 29;397(10289):2098-2110. doi: 10.1016/S0140-6736(21)00392-5. PMID 34062144
- [Background] Kosek E, Cohen M, Baron R, Gebhart GF, Mico JA, Rice ASC, Rief W, Sluka AK. Do we need a third mechanistic descriptor for chronic pain states? Pain. 2016 Jul;157(7):1382-1386. doi: 10.1097/j.pain.0000000000000507. No abstract available. PMID 26835783
- [Background] Gooren LJ, Sungkaew T, Giltay EJ, Guadamuz TE. Cross-sex hormone use, functional health and mental well-being among transgender men (Toms) and Transgender Women (Kathoeys) in Thailand. Cult Health Sex. 2015;17(1):92-103. doi: 10.1080/13691058.2014.950982. Epub 2014 Oct 1. PMID 25270637
- [Background] Motmans J, Meier P, Ponnet K, T'Sjoen G. Female and male transgender quality of life: socioeconomic and medical differences. J Sex Med. 2012 Mar;9(3):743-50. doi: 10.1111/j.1743-6109.2011.02569.x. Epub 2011 Dec 21. PMID 22188877
- [Background] Valashany BT, Janghorbani M. Quality of life of men and women with gender identity disorder. Health Qual Life Outcomes. 2018 Aug 20;16(1):167. doi: 10.1186/s12955-018-0995-7. PMID 30126432
- [Background] Gorin-Lazard A, Baumstarck K, Boyer L, Maquigneau A, Gebleux S, Penochet JC, Pringuey D, Albarel F, Morange I, Loundou A, Berbis J, Auquier P, Lancon C, Bonierbale M. Is hormonal therapy associated with better quality of life in transsexuals? A cross-sectional study. J Sex Med. 2012 Feb;9(2):531-41. doi: 10.1111/j.1743-6109.2011.02564.x. Epub 2011 Dec 6. PMID 22145968
- [Background] Weyers S, Elaut E, De Sutter P, Gerris J, T'Sjoen G, Heylens G, De Cuypere G, Verstraelen H. Long-term assessment of the physical, mental, and sexual health among transsexual women. J Sex Med. 2009 Mar;6(3):752-60. doi: 10.1111/j.1743-6109.2008.01082.x. Epub 2008 Nov 17. PMID 19040622
- [Background] Levit D, Yaish I, Shtrozberg S, Aloush V, Greenman Y, Ablin JN. Pain and transition: evaluating fibromyalgia in transgender individuals. Clin Exp Rheumatol. 2021 May-Jun;39 Suppl 130(3):27-32. doi: 10.55563/clinexprheumatol/pq0qp6. Epub 2021 Jan 13. PMID 33506751
- [Background] Athnaiel O, Cantillo S, Paredes S, Knezevic NN. The Role of Sex Hormones in Pain-Related Conditions. Int J Mol Sci. 2023 Jan 18;24(3):1866. doi: 10.3390/ijms24031866. PMID 36768188
- [Background] Seelman KL, Young SR, Tesene M, Alvarez-Hernandez LR, Kattari L. A Comparison of Health Disparities among Transgender Adults in Colorado (USA) by Race and Income. Int J Transgend. 2017;18(2):199-214. doi: 10.1080/15532739.2016.1252300. Epub 2016 Nov 22. PMID 33132785
- [Background] Aloisi AM, Bachiocco V, Costantino A, Stefani R, Ceccarelli I, Bertaccini A, Meriggiola MC. Cross-sex hormone administration changes pain in transsexual women and men. Pain. 2007 Nov;132 Suppl 1:S60-S67. doi: 10.1016/j.pain.2007.02.006. Epub 2007 Mar 26. PMID 17379410
- [Background] Dragon CN, Guerino P, Ewald E, Laffan AM. Transgender Medicare Beneficiaries and Chronic Conditions: Exploring Fee-for-Service Claims Data. LGBT Health. 2017 Dec;4(6):404-411. doi: 10.1089/lgbt.2016.0208. Epub 2017 Nov 10. PMID 29125908
- [Background] Irwig MS. Testosterone therapy for transgender men. Lancet Diabetes Endocrinol. 2017 Apr;5(4):301-311. doi: 10.1016/S2213-8587(16)00036-X. Epub 2016 Apr 12. PMID 27084565
- [Background] Tangpricha V, den Heijer M. Oestrogen and anti-androgen therapy for transgender women. Lancet Diabetes Endocrinol. 2017 Apr;5(4):291-300. doi: 10.1016/S2213-8587(16)30319-9. Epub 2016 Dec 2. PMID 27916515
- [Background] Craft RM, Mogil JS, Aloisi AM. Sex differences in pain and analgesia: the role of gonadal hormones. Eur J Pain. 2004 Oct;8(5):397-411. doi: 10.1016/j.ejpain.2004.01.003. PMID 15324772
- [Background] Li H, Neubauer SA, Hayes DL. Follow-up of a minute ventilation rate adaptive pacemaker. Pacing Clin Electrophysiol. 1992 Nov;15(11 Pt 2):1826-9. doi: 10.1111/j.1540-8159.1992.tb02976.x. PMID 1279555
- [Background] Wiesenfeld-Hallin Z. Sex differences in pain perception. Gend Med. 2005 Sep;2(3):137-45. doi: 10.1016/s1550-8579(05)80042-7. PMID 16290886
- [Background] LeResche L, Mancl LA, Drangsholt MT, Saunders K, Von Korff M. Relationship of pain and symptoms to pubertal development in adolescents. Pain. 2005 Nov;118(1-2):201-9. doi: 10.1016/j.pain.2005.08.011. Epub 2005 Oct 5. PMID 16213087